CLINICAL TRIAL: NCT03175224
Title: Phase 1 / 2 Multicenter Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of APL-101 in Subjects With Non-Small Cell Lung Cancer With c-Met EXON 14 Skip Mutations and c-Met Dysregulation Advanced Solid Tumors
Brief Title: APL-101 Study of Subjects With NSCLC With c-Met EXON 14 Skip Mutations and c-Met Dysregulation Advanced Solid Tumors
Acronym: SPARTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apollomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-101-01
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Advanced Cancer; Renal Cancer; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; NSCLC; Lung Cancer; Brain Tumor; Glioblastoma Multiforme; EGFR Gene Mutation; MET Amplification; HGF; Thyroid Cancer; Pancreatic Cancer; Colon Cancer; MET Alteration; MET Fusion; Exon 14 Skipping
Keywords: Advanced Solid Tumor; Relapsed Solid Tumor; Recurrent Solid Tumor; cMet exon 14 skipping; cMet fusion; GBM; HGF; EGFR positive
MeSH Terms: conditions — Kidney Neoplasms; Stomach Neoplasms; Lung Neoplasms; Brain Neoplasms; Glioblastoma; Thyroid Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- NSCLC Exon 14 Skip Treatment Naive (Experimental): Cohort A-1: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- NSCLC Exon 14 Skip Previously Treated (Experimental): Cohort A-2: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- NSCLC Exon 14 MET Inhibitor Experienced (Experimental): Cohort B: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- Basket of tumor types MET amplification except for primary CNS tumors (Experimental): Cohort C: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- NSCLC MET amplification and EGFR wild-type (Experimental): Cohort C-1: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- EGFR positive NSCLC MET amplification as an acquired resistance (Experimental): Cohort C-2: APL-101 Oral Capsules + Standard of Care EGFR Inhibitor
  Interventions: Drug: APL-101 Oral Capsules
- Basket of solid tumor with MET gene fusions except for primary CNS tumors (Experimental): Cohort D: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- Primary CNS tumors with MET alterations (Experimental): Cohort E: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules
- Basket of tumor types wild-type MET with over-expression of HGF and MET (Experimental): Cohort F: APL-101 Oral Capsules
  Interventions: Drug: APL-101 Oral Capsules

INTERVENTIONS:
Drug: APL-101 Oral Capsules — Subjects will receive APL-101 capsules BID for oral administration.
  Other Names: PLB-1001; CBI-3103; Bozitinib; CBT-101; Vebreltinib

SUMMARY:
To assess:

* efficacy of APL-101 as monotherapy for the treatment of NSCLC harboring MET Exon 14 skipping mutations, NSCLC harboring MET amplification, solid tumors harboring MET amplification, solid tumors harboring MET fusion, primary CNS tumors harboring MET alterations, solid tumors harboring wild-type MET with overexpression of HGF and MET
* efficacy of APL-101 as an add-on therapy to EGFR inhibitor for the treatment of NSCLC harboring EGFR activating mutations and developed acquired resistance with MET amplification and disease progression after documented CR or PR with 1st line EGFR inhibitors (EGFR-I)

DETAILED DESCRIPTION:
Phase 1 (lead-in stage of this study) enrollment has been completed.

In this Phase 2 study, efficacy, safety, and tolerability will be assessed in the following cohorts:

* Cohort A-1: NSCLC EXON 14 skip mutation, previously untreated, MET inhibitor naive (c-Met naïve, 1L)
* Cohort A-2: NSCLC EXON 14 skip mutation, previously treated with ≤ 3 prior lines in unresectable or metastatic setting, MET inhibitor naive (c-Met naïve, 2/3L)
* Cohort B: NSCLC EXON 14 skip mutation, previously treated with ≤ 3 prior lines in unresectable or metastatic setting, MET inhibitor experienced (c-Met experienced; progressed on prior c-Met inhibitor)
* Cohort C: basket of tumor types (e.g., NSCLC, upper gastrointestinal [GI], colorectal, hepatobiliary cancer) harboring MET amplification except for primary CNS tumors, previously treated or previously untreated but refused standard treatment, or if treatment was unavailable or unfeasible (≤ 3 prior lines in unresectable or metastatic setting), MET inhibitor naïve
* Cohort C-1: NSCLC harboring MET amplification and wild-type epidermal growth factor receptor (EGFR), previously treated; or untreated but refused standard treatment, or if treatment was unavailable or unfeasible (≤ 3 prior lines in unresectable or metastatic setting), MET inhibitor naïve
* Cohort C-2: EGFR positive NSCLC harboring MET amplification as an acquired resistance, documented response with first-line EGFR-Inhibitor (PR or CR per RECIST ≥ 12 weeks), radiological documentation of disease progression per RECIST on first-line EGFR inhibitor therapy, MET inhibitor naïve
* Cohort D: basket of tumor types except for primary CNS tumors harboring MET gene fusions (e.g., NSCLC, upper GI, colorectal, hepatobiliary cancer), previously treated; or previously untreated but refused standard treatment, or if treatment was unavailable or unfeasible (≤ 3 prior lines in unresectable or metastatic setting), MET inhibitor naïve
* Cohort E: primary CNS tumors with MET alterations (single or co-occurred MET fusion including PTPRZ1-MET [ZM] fusion, MET Exon 14 skipping mutation, or MET amplification), previously treated or previously untreated but refused standard treatment, or if treatment was unavailable or unfeasible (≤ 3 prior lines), MET inhibitor naïve
* Cohort F: basket of tumor types harboring wild-type MET with over-expression of HGF and MET (e.g., NSCLC, upper GI, colorectal, hepatobiliary cancer or primary CNS tumors), previously treated; or previously untreated but refused standard treatment, or if treatment was unavailable or unfeasible (≤ 3 prior lines in unresectable or metastatic setting), MET inhibitor naïve

ELIGIBILITY:
Major Inclusion Criteria:

1. Men and women 18 years of age or older.
2. 9 cohorts will be enrolled:

   * Cohort A1 / Exon 14 NSCLC MET inhibitor naive in first line: Histologically or cytologically confirmed NSCLC with Exon 14 skipping mutations; all histologies; unresectable or metastatic disease (Stage 3b/4); treatment-naive subjects in first line; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort A2 / Exon 14 NSCLC - MET inhibitor naïve: Histologically or cytologically confirmed NSCLC with Exon 14 skipping mutations; all histologies; unresectable or metastatic disease (Stage 3b/4); pretreated subjects refractory to or intolerant of standard therapies with no more than three lines of prior therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort B / Exon 14 NSCLC MET inhibitor experienced: ENROLLMENT COMPLETED
   * Cohort C / MET amplification basket tumor types excluding primary CNS tumors: Any solid tumor type regardless of histology excluding primary CNS tumors, with MET amplification; unresectable or metastatic disease, refractory to or intolerant of standard therapies, or refused standard therapies, or if therapy was unavailable or unfeasible, with no more than 3 prior lines of therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort C1 / MET amplification and wild-type EGFR NSCLC: NSCLC regardless of histology, harboring MET amplification and wild-type EGFR; unresectable or metastatic disease, previously untreated or treated with no more than 3 prior lines of therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort C2 / EGFR positive NSCLC with acquired MET amplification (APL-101 Add-on Therapy): Unresectable or metastatic NSCLC regardless of histology, harboring EGFR activating mutations with acquired MET-Amplification as resistance mechanism to the EGFR-I; developed resistance to first-line EGFR-inhibitor therapy after an initial response (documented PR for at least 12 weeks); radiological documentation of disease progression per RECIST on first-line EGFR inhibitor therapy; currently on an EGFR-inhibitor therapy and agrees to receive APL-101 as an add-on therapy during the study; no history of interstitial lung disease (ILD)/pneumonitis, Grade ≥3 liver toxicity or QT prolongation with EGFR-I therapy; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort D / MET fusion basket tumor types excluding primary CNS tumors: any solid tumor type regardless of histology excluding primary CNS tumors; unresectable or metastatic disease, refractory to or intolerant of standard therapies, or refused standard therapies, or if therapy was unavailable or unfeasible, with no more than 3 prior lines of therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
   * Cohort E / Primary CNS tumors with MET alterations: subjects with primary CNS tumors who meet inclusion criteria of MET dysregulations defined as single or co-occurred MET fusion including PTPRZ1-MET (ZM) fusion, MET Exon 14 skipping mutations, or MET amplification; refractory to or intolerant of standard therapies, or refused standard therapies, or if therapy was unavailable or unfeasible, with no more than 3 prior lines of therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations; neurological symptoms controlled on a stable/decreasing dose of steroids for at least 2 weeks before C1D1
   * Cohort F / Basket tumor types harboring wild-type MET with over-expression of HGF and MET: any solid tumor type regardless of histology harboring wild-type MET with overexpression of HGF and MET; Unresectable or metastatic disease, refractory to or intolerant of standard therapies, or refused standard therapies, or if therapy was unavailable or unfeasible, with no more than 3 prior lines of therapy in the unresectable or metastatic setting; not received any MET inhibitor and no known MET kinase inhibitor resistance mutations
3. Treated or untreated asymptomatic parenchymal CNS disease or leptomeningeal disease is allowed.
4. Presence of ≥1 measurable lesion (scan done ≤28 days of C1D1) to serve as target lesion according to relevant criteria
5. ECOG performance status of 0-1. For subjects with primary CNS tumors, KPS score ≥70.
6. Acceptable organ function
7. For all prior anticancer treatment, a duration of 30 days or 5 half-lives of the agents used, whichever is shorter, must have elapsed, and any encountered toxicity must have resolved to levels meeting all the other eligibility criteria prior to the first dose of study treatment. Palliative radiotherapy to non-target lesions should be completed within 2 weeks prior to APL-101 administration.
8. Adequate cardiac function
9. Women of child-bearing potential must have a negative serum or Beta-hCG at screening or evidence of surgical sterility or evidence of post-menopausal status
10. No planned major surgery within 4 weeks of first dose of APL-101
11. Expected survival (life expectancy) ≥ 3 months from C1D1
12. Provision of sample; e.g. archival or a fresh tumor biopsy sample (if safe and feasible) either from the primary or a metastatic site) or liquid biopsy sample (if tumor tissue is insufficient or lacking, and approved by the sponsor) is required for prospective central lab confirmation for study entry (subjects with previously confirmed molecular status by the Sponsor designated central lab or FDA approved NGS based MET testing may be exempted, subjected to Sponsor approval.

Major Exclusion Criteria:

1. Hypersensitivity to APL-101, excipients of the drug product, or other components of the study treatment regimen.
2. Known actionable mutation/gene rearrangement of EGFR (except for NSCLC subjects in Cohort C and C-2), ALK, ROS1, RET, NTRK, KRAS, and BRAF.
3. Use or intended use of any other investigational product, including herbal medications, through Study Treatment Termination.
4. Active uncontrolled systemic bacterial, viral, or fungal infection or clinically significant, active disease process, which in the opinion of the investigator makes the risk: benefit unfavorable for the participation of the trial.
5. Life-threatening illness, significant organ system dysfunction or comorbid conditions, or other reasons that, in the investigator's opinion, could compromise the subject's safety or the integrity of the study outcomes, or interfere with the absorption or metabolism of APL-101.
6. Unstable angina or myocardial infarction within 1 year prior to first dose of APL-101, symptomatic or unstable arrhythmia requiring medical therapy, history of congenital prolonged QT syndrome, prolonged QT interval corrected by Fridericia formula (QTcF) at screening, or concurrent treatment with a medication that is a known risk for prolonging the QT interval. Chronic controlled atrial fibrillation is not excluded.
7. Historical seropositive results consistent with active infection for hepatitis C virus (HCV) or hepatitis B virus (HBV) with high viral loads not actively managed with antiviral therapy and human immunodeficiency virus (HIV) positive subjects who are not clinically stable or controlled on their medication (asymptomatic subjects with CD4+ T-cell (CD4+) counts ≥ 350 cells/μL and have not had an opportunistic infection within the past 12 months prior to first dose of APL-101 would be eligible for study entry. If history is unclear, relevant test(s) at Screening will be required to confirm eligibility.
8. Known significant mental illness or other conditions such as active alcohol or other substance abuse that, in the opinion of the investigator, predisposes the subject to high risk of noncompliance with the protocol treatment or assessments.
9. Unable to swallow orally administered medication whole.
10. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption
11. Women who are breastfeeding
12. History of another malignancy within 3 years prior to C1D1. A subject with the following malignancies is allowed if considered cured or unlikely to recur within 3 years:

    1. Carcinoma of the skin without melanomatous features.
    2. Curatively treated cervical carcinoma in situ.
    3. Bladder tumors considered superficial such as noninvasive (T1a) and carcinoma in situ (T1s), thyroid papillary cancer with prior treatment, prostate cancer which has been surgically or medically treated and not likely to recur within 3 years.
13. Subjects who are unable or unwilling to discontinue excluded medications (drugs with known QTc risk and known strong cytochrome P450 [CYP]3A4 inducer and/or strong inhibitors) for at least 5 half-lives prior to first dose of study drug. Subjects may qualify if such medication(s) can be safely replaced with alternate medications with less risk of drug-drug interaction.
14. Subjects with active COVID-19 infection.
15. Symptomatic and/or neurologically unstable CNS metastases, or who require an increase in steroid dose to control CNS disease. Subjects who have been receiving a stable steroid dose for at least 2 weeks prior to C1D1 may be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR = CR + PR) per IRC committee (BIRC) based on RECIST v1.1 (or relevant criteria per tumor type) | From time of informed consent signature through completion of treatment (1 cycle = 28 days) or progression
  Anti-tumor activity per RECIST v1.1, RANO criteria for CNS tumors, or relevant evaluation criteria per tumor type.

SECONDARY OUTCOMES:
Median duration of response (DOR) per IRC. | Approximately 2 years
  DOR per RECIST v1.1 criteria, RANO criteria for CNS tumors, or relevant evaluation criteria per tumor type.
ORR per investigator assessment based on RECIST v1.1. | Approximately 2 years
  ORR per RECIST v1.1 or relevant evaluation criteria per tumor type.
Median DOR per investigator assessment. | Approximately 2 years
  DOR per RECIST v1.1, RANO criteria for CNS tumors, or relevant evaluation criteria per tumor type.
Antitumor activity by clinical benefit rate (CR + PR + SD ≥ 4 cycles) based on RECIST v1.1, RANO criteria for CNS tumors, or other relevant criteria per tumor type Median time to progression (TTP). | Approximately 2 years
  Benefit rate per RECIST v1.1, RANO criteria for CNS tumors, or relevant evaluation criteria per tumor type.
Median time to progression (TTP). | Approximately 2 years
  TTP per RECIST v1.1 or relevant evaluation criteria per tumor type.
Progression Free Survival (PFS) and overall survival (OS) at 6, 12, 18 and 24 months | Approximately 3 years
  PFS and OS per RECIST v1.1 or relevant evaluation criteria per tumor type.

CONTACTS AND LOCATIONS:
Overall Officials: Mythili Sangem, Study Director — Apollomics Inc.
Locations (35):
- United States (6):
  - Cedars-Sinai Medical Center - Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Moffitt, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
- St Vincents Hospital Melbourne, Melbourne, Australia
- Canada (4):
  - Cross Cancer Institute, Edmonton
  - McGill University Health Center - Research Institute, Montreal
  - Princess Margaret Hospital, Toronto
  - Cancer Care Manitoba, Winnipeg
- France (5):
  - CHRU de Brest - Hôpital Morvan, Brest
  - Centre Leon Berard, Lyon
  - Centre d'Essais Precoces en Cancerologie de Marseille, Marseille
  - Hopital Bichat - Claude Bernard - AP-HP, Paris
  - Gustave Roussy, Villejuif
- Hungary (2):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Oncologico Veneto-I.R.C.C.S. - Ospedale Busonera, Padua
- Private Medical Institution Euromedservice, Saint Petersburg, Russia
- National Cancer Centre Singapore, Singapore, Singapore
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto Valenciano de Oncologia, Valencia
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (3):
  - University College London Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital - Surrey, Surrey Quays

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Apollomics, Inc. website — https://www.apollomicsinc.com